CLINICAL TRIAL: NCT05895279
Title: Minority Prostate Cancer (MiCaP) Phase III (Aim 3): Assessment of Research Digest Impact
Brief Title: Assessment of Research Digest Impact for Minority with Prostate Cancer, MiCAP Phase III Study
Acronym: MiCaP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-006715; NCI-2022-09906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-006715 (Other: Mayo Clinic Institutional Review Board); MiCaP (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2023-05-17; First posted 2023-06-08 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MiCaP Research Digest Video Group (Experimental): Participants watch MiCaP Research Digest video on study. Participants complete a survey throughout the trial.
  Interventions: Other: Media Intervention; Other: Survey Administration
- Alternate Video Group (Active Comparator): Participants watch an alternative video on study. Participants complete a survey throughout the trial.
  Interventions: Other: Media Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Media Intervention — Watch MiCaP Research Digest video
  Arms: MiCaP Research Digest Video Group
Other: Media Intervention — Watch alternate video
  Arms: Alternate Video Group
Other: Survey Administration — Complete survey

SUMMARY:
This phase III trial determines how well the Minority Prostate Cancer (MiCaP) Research Digest works in providing information to black men about the latest prostate cancer research. MiCaP Research Digest may be an effective method to help people learn about prostate cancer.This goal of this trial is to create educational programming that helps Black men make informed decisions about their prostate healthcare since Black men are diagnosed with prostate cancer more than any other race or ethnicity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop a research dissemination program, the Minority Prostate Cancer (MiCaP) Research Digest, which will spread information about CaP scientific discoveries, evidence-based interventions, and open clinical trials instantly among black males (BM).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants watch MiCaP Research Digest video on study. Participants complete a survey throughout the trial.

ARM II: Participants watch an alternative video on study. Participants complete a survey throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a Black male
* Between the ages of 35 and 70
* For virtual data collection, have access to the internet and Zoom (if joining study online)
* For virtual data collection, reside anywhere in the U.S.
* For in-person data collection, reside in one of the nine (9) catchment areas of the Mayo Clinic Cancer Center: Baker, Duval, Nassau, Clay, St. John's, Putnam, Flagler, Volusia and Brevard

Exclusion Criteria:

* Identify as a race or ethnicity that is not Black
* Identify as female
* Be younger than age 35 and older than age 70
* Lack access to internet and Zoom (if joining study online)

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in perception of access to medical services and general health | Baseline, 1 hour after video intervention
  Using the Minority Prostate Cancer (MiCaP) survey developed for this study, participants are asked 10 questions regarding access to medical services and general health with a yes/no response.
Change in perception in participation with clinical trials about prostate cancer | Baseline, 1 hour after video intervention
  Using the Minority Prostate Cancer (MiCaP) survey developed for this study, participants are asked 10 questions regarding views on participating in clinical trials about prostate cancer with a yes/no response.
Change in perception of familiarity with prostate cancer research | Baseline, 1 hour after video intervention
  Using the Minority Prostate Cancer (MiCaP) survey developed for this study, participants are asked 5 questions regarding views on participating in clinical trials about prostate cancer with a true/false/don't know response.
Change in perception of familiarity with a research study protocol | Baseline, 1 hour after video intervention
  Using the Minority Prostate Cancer (MiCaP) survey developed for this study, participants are asked 5 questions regarding information about a study protocol with a true/false/don't know response.

CONTACTS AND LOCATIONS:
Overall Officials: Folakemi T. Odedina, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials